CLINICAL TRIAL: NCT04944498
Title: Modified Tarsorrhaphy vs Gold Weight Implant Technique for Paralytic Lagophthalmos Treatment in Leprosy Patients: a Randomized Clinical Trial
Brief Title: Modified Tarsorrhaphy vs Gold Weight Implant for Paralytic Lagophthalmos in Leprosy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yunia Irawati (Other)
Responsible Party: Sponsor-Investigator, Yunia Irawati, Principal Investigator, Gadjah Mada University
Organization: Gadjah Mada University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KE/FK/0525/EC/2019
Record Dates: First submitted 2021-06-04; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Paralytic Lagophthalmos; Leprosy--Patients
Keywords: Hansen Disease; Leprosy; Paralytic lagophthalmos; Surgical intervention
MeSH Terms: conditions — Lagophthalmos; Leprosy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Treatment received by patients was randomized by research team members. The investigator as the oculoplastic surgeon (YI) acknowledged the treatment assigned to each patient based on randomization. Outcomes were measured by other oculoplastic surgeons with equal clinical experiences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients who received surgery with modified tarsorrhaphy technique
  Interventions: Procedure: Modified Tarsorrhaphy
- Control group (Active Comparator): Patients who received surgery with gold weight implant technique
  Interventions: Procedure: Gold Weight Implant

INTERVENTIONS:
Procedure: Modified Tarsorrhaphy — A combination of levator recess, lateral tarsorrhaphy of 10 mm, and lateral canthopexy/lateral tarsal strip
  Arms: Intervention Group
Procedure: Gold Weight Implant — Installation of 1,5 gram gold weight implant above tarsal plate and underneath levator recess
  Arms: Control group

SUMMARY:
This study aims to compare the effectivity and efficiency of Modified Tarsorrhaphy (MT) technique and Gold Weight Implant (GWI) technique as a surgical treatment of paralytic lagophthalmos in leprosy patients. The hypothesis is that MT technique is more effective and more efficient than GWI technique. This study used PROBE (Prospective Randomized Open-label Blinded-Endpoint) clinical trial. Samples consisted of 14 eyes in MT group and 13 eyes in GWI group as the control group. This study was conducted in 3 hospitals in Indonesia and the patients were observed in 1 year period.

ELIGIBILITY:
Inclusion Criteria:

* paucibacillary (PB) or multibacillary (MB) type leprosy patient with unilateral/bilateral lagophthalmos who had not undergone eyelid reconstruction
* patient aged 18 years old or older who could be performed surgery with local anesthesia

Exclusion Criteria:

* patient with acute leprosy reaction (<6 months) and in steroid medication
* patient with eyelid laxity >8 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2021-04-04 (Actual)

PRIMARY OUTCOMES:
Lagophthalmos distance without pressure | Pre-operative
  Eyelid margin distance in central, nasal, and temporal area measured in millimeters
Lagophthalmos distance without pressure | 1 day post-operative
  Eyelid margin distance in central, nasal, and temporal area measured in millimeters
Lagophthalmos distance without pressure | 7 day post-operative
  Eyelid margin distance in central, nasal, and temporal area measured in millimeters
Lagophthalmos distance without pressure | 1 month post-operative
  Eyelid margin distance in central, nasal, and temporal area measured in millimeters
Lagophthalmos distance without pressure | 3 months post-operative
  Eyelid margin distance in central, nasal, and temporal area measured in millimeters
Lagophthalmos distance without pressure | 1 year post-operative
  Eyelid margin distance in central, nasal, and temporal area measured in millimeters
Lagophthalmos distance with gentle pressure | Pre-operative
  Eyelid margin distance in central, nasal, and temporal area measured in millimeters after applying minimal pressure on upper eyelid
Lagophthalmos distance with gentle pressure | 1 day post-operative
  Eyelid margin distance in central, nasal, and temporal area measured in millimeters after applying minimal pressure on upper eyelid
Lagophthalmos distance with gentle pressure | 7 day post-operative
  Eyelid margin distance in central, nasal, and temporal area measured in millimeters after applying minimal pressure on upper eyelid
Lagophthalmos distance with gentle pressure | 1 month post-operative
  Eyelid margin distance in central, nasal, and temporal area measured in millimeters after applying minimal pressure on upper eyelid
Lagophthalmos distance with gentle pressure | 3 months post-operative
  Eyelid margin distance in central, nasal, and temporal area measured in millimeters after applying minimal pressure on upper eyelid
Lagophthalmos distance with gentle pressure | 1 year post-operative
  Eyelid margin distance in central, nasal, and temporal area measured in millimeters after applying minimal pressure on upper eyelid
OSDI (Ocular Surface Disease Index) | Pre-operative
  Questionnaire assessing subjective dry eyes symptoms
OSDI (Ocular Surface Disease Index) | 1 day post-operative
  Questionnaire assessing subjective dry eyes symptoms
OSDI (Ocular Surface Disease Index) | 7 day post-operative
  Questionnaire assessing subjective dry eyes symptoms
OSDI (Ocular Surface Disease Index) | 1 month post-operative
  Questionnaire assessing subjective dry eyes symptoms
OSDI (Ocular Surface Disease Index) | 3 month post-operative
  Questionnaire assessing subjective dry eyes symptoms
OSDI (Ocular Surface Disease Index) | 1 year post-operative
  Questionnaire assessing subjective dry eyes symptoms
TBUT (Tear Break-Up Time) | Pre-operative
  Examination of tear break up time with fluorescein dye assessed with cobalt blue light from slit lamp
TBUT (Tear Break-Up Time) | 1 day post-operative
  Examination of tear break up time with fluorescein dye assessed with cobalt blue light from slit lamp
TBUT (Tear Break-Up Time) | 7 day post-operative
  Examination of tear break up time with fluorescein dye assessed with cobalt blue light from slit lamp
TBUT (Tear Break-Up Time) | 1 month post-operative
  Examination of tear break up time with fluorescein dye assessed with cobalt blue light from slit lamp
TBUT (Tear Break-Up Time) | 3 months post-operative
  Examination of tear break up time with fluorescein dye assessed with cobalt blue light from slit lamp
Schirmer test without anesthesia | Pre-operative
  Tear film excretion examined using Whatman filter paper without anesthesia
Schirmer test without anesthesia | 1 day post-operative
  Tear film excretion examined using Whatman filter paper without anesthesia
Schirmer test without anesthesia | 7 day post-operative
  Tear film excretion examined using Whatman filter paper without anesthesia
Schirmer test without anesthesia | 1 month post-operative
  Tear film excretion examined using Whatman filter paper without anesthesia
Schirmer test without anesthesia | 3 months post-operative
  Tear film excretion examined using Whatman filter paper without anesthesia
Schirmer test without anesthesia | 1 year post-operative
  Tear film excretion examined using Whatman filter paper without anesthesia
Schirmer test with anesthesia | Pre-operative
  Tear film excretion examined using Whatman filter paper with anesthesia prior to examination
Schirmer test with anesthesia | 1 day post-operative
  Tear film excretion examined using Whatman filter paper with anesthesia prior to examination
Schirmer test with anesthesia | 7 day post-operative
  Tear film excretion examined using Whatman filter paper with anesthesia prior to examination
Schirmer test with anesthesia | 1 month post-operative
  Tear film excretion examined using Whatman filter paper with anesthesia prior to examination
Schirmer test with anesthesia | 3 months post-operative
  Tear film excretion examined using Whatman filter paper with anesthesia prior to examination
Schirmer test with anesthesia | 1 year post-operative
  Tear film excretion examined using Whatman filter paper with anesthesia prior to examination
Epitheliopathy | Pre-operative
  Epitheliopathy occurence, assessed with fluorescent dye and observed with cobalt blue light filter of slit lamp
Epitheliopathy | 1 day post-operative
  Epitheliopathy occurence, assessed with fluorescent dye and observed with cobalt blue light filter of slit lamp
Epitheliopathy | 7 day post-operative
  Epitheliopathy occurence, assessed with fluorescent dye and observed with cobalt blue light filter of slit lamp
Epitheliopathy | 1 month post-operative
  Epitheliopathy occurence, assessed with fluorescent dye and observed with cobalt blue light filter of slit lamp
Epitheliopathy | 3 months post-operative
  Epitheliopathy occurence, assessed with fluorescent dye and observed with cobalt blue light filter of slit lamp
Corneal exposure | Pre-operative
  Exposed distance of cornea when the eye was closed
Corneal exposure | 1 day post-operative
  Exposed distance of cornea when the eye was closed
Corneal exposure | 7 day post-operative
  Exposed distance of cornea when the eye was closed
Corneal exposure | 1 month post-operative
  Exposed distance of cornea when the eye was closed
Corneal exposure | 3 months post-operative
  Exposed distance of cornea when the eye was closed
Corneal sensibility | Pre-operative
  Sensibility measured in millimeters by using Luneau Cohcet-Bonnet Aesthesiometer
Corneal sensibility | 1 day post-operative
  Sensibility measured in millimeters by using Luneau Cohcet-Bonnet Aesthesiometer
Corneal sensibility | 7 day post-operative
  Sensibility measured in millimeters by using Luneau Cohcet-Bonnet Aesthesiometer
Corneal sensibility | 1 month post-operative
  Sensibility measured in millimeters by using Luneau Cohcet-Bonnet Aesthesiometer
Corneal sensibility | 3 months post-operative
  Sensibility measured in millimeters by using Luneau Cohcet-Bonnet Aesthesiometer
Complication | intraoperative
  Complication during surgery and after surgery
Complication | 1 day post-operative
  Complication during surgery and after surgery
Complication | 7 day post-operative
  Complication during surgery and after surgery
Complication | 1 month post-operative
  Complication during surgery and after surgery
Complication | 3 months post-operative
  Complication during surgery and after surgery
Complication | 1 year post-operative
  Complication during surgery and after surgery
Duration | Intraoperative
  Duration of surgery
Cost | 1 year post-operative
  Cost of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yunia Irawati, Ophthalmologist Consultant, Principal Investigator — Indonesia University
Locations (3):
- Indonesia (3):
  - Jakarta Eye Center Hospitals and Clinics, Jakarta, DKI Jakarta
  - dr. Cipto Mangunkusumo Kirana Eye Hospital, Jakarta Pusat, DKI Jakarta
  - dr. Tadjuddin Chalid General Hospital, Makassar, South Sulawesi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pereira MV, Gloria AL. Lagophthalmos. Semin Ophthalmol. 2010 May;25(3):72-8. doi: 10.3109/08820538.2010.488578. PMID 20590416
- [Background] El Toukhy E. Gold weight implants in the management of lagophthalmos in leprosy patients. Lepr Rev. 2010 Mar;81(1):79-81. PMID 20496572
- [Background] Daniel E, Koshy S, Joseph GA, Rao PS. Ocular complications in incident relapsed borderline lepromatous and lepromatous leprosy patients in south India. Indian J Ophthalmol. 2003 Jun;51(2):155-9. PMID 12831146
- [Background] Nemet AY. Augmentation of lateral tarsorrhaphy in lagophthalmos. Orbit. 2014 Aug;33(4):289-91. doi: 10.3109/01676830.2014.894537. Epub 2014 Apr 30. PMID 24786615
- [Background] Aggarwal E, Naik MN, Honavar SG. Effectiveness of the gold weight trial procedure in predicting the ideal weight for lid loading in facial palsy: a prospective study. Am J Ophthalmol. 2007 Jun;143(6):1009-1012. doi: 10.1016/j.ajo.2007.03.026. Epub 2007 Apr 20. PMID 17449001
- [Background] Hontanilla B. Weight measurement of upper eyelid gold implants for lagophthalmos in facial paralysis. Plast Reconstr Surg. 2001 Nov;108(6):1539-43. doi: 10.1097/00006534-200111000-00016. PMID 11711925
- [Background] Lamba PA, Srinivasan R, Rohatgi J. Surgical management in ocular leprosy. Indian J Ophthalmol. 1987 May-Jun;35(3):153-7. No abstract available. PMID 3507412
- [Background] Koshy S, Daniel E, Kurian N, Yovan P. Pathogenesis of dry eye in leprosy and tear functions. Int J Lepr Other Mycobact Dis. 2001 Sep;69(3):215-8. PMID 11875765
- [Background] Li W, Yeh TN, Leung T, Yuen T, Lerma M, Lin MC. The Relationship of Lid Wiper Epitheliopathy to Ocular Surface Signs and Symptoms. Invest Ophthalmol Vis Sci. 2018 Apr 1;59(5):1878-1887. doi: 10.1167/iovs.17-23639. PMID 29677348
- [Background] Harrisberg BP, Singh RP, Croxson GR, Taylor RF, McCluskey PJ. Long-term outcome of gold eyelid weights in patients with facial nerve palsy. Otol Neurotol. 2001 May;22(3):397-400. doi: 10.1097/00129492-200105000-00022. PMID 11347647
- [Background] Hieselaar LC, Hogeweg M, de Vries CL. Corneal sensitivity in patients with leprosy and in controls. Br J Ophthalmol. 1995 Nov;79(11):993-5. doi: 10.1136/bjo.79.11.993. PMID 8534670
- [Background] Karacorlu MA, Cakiner T, Saylan T. Corneal sensitivity and correlations between decreased sensitivity and anterior segment pathology in ocular leprosy. Br J Ophthalmol. 1991 Feb;75(2):117-9. doi: 10.1136/bjo.75.2.117. PMID 1995039